CLINICAL TRIAL: NCT01508299
Title: Skin Prick Test for the Diagnosis of Food Allergy- a Comparison of Different Commercial Extracts and Raw Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Arnon Goldberg, Professor, Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: crufood1
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Food Allergy
Keywords: skin test; raw food; commercial extract
MeSH Terms: conditions — Food Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- raw food skin test (Experimental): skin test with the suspected raw food
  Interventions: Procedure: skin test

INTERVENTIONS:
Procedure: skin test — skin test with the Suspected raw food

SUMMARY:
Immediate food allergy is , sometimes , a life threatening situation . Diagnosis is done by skin prick test with commercial extracts. Nevertheless, some of the extracts are not optimal and reproduce false negative results (no allergy) in patients with history highly suggestive of allergic reaction. The aim of this study is to compare the reproducibility of different commercial extracts and raw food in patients with convincing history of acute allergic symptoms related to food .

ELIGIBILITY:
Inclusion Criteria:

* Suspected immediate allergic reaction to food

Exclusion Criteria:none

Ages: 1 Month to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
correlation between the results of skin test with commercial extracts and raw food | immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy and clinical immunology unit , Meir hospital, Kfar Saba, Israel, Israel